CLINICAL TRIAL: NCT07168135
Title: Effect of Discontinuing Propofol Anesthesia After Cecal Intubation on Patient's Psychomotor Recovery Following Colonoscopy: A Prospective Two-Arm Parallel Randomized Double-Blind Interventional Controlled Trial
Brief Title: Effect of Discontinuing Propofol After Cecal Intubation on Patient's Psychomotor Recovery Following Colonoscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ala'a Sharara, MD, Professor of Gastroenterology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BIO-2024-0344
Record Dates: First submitted 2025-08-25; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Procedural Sedation; Colonoscopy; Cecal Intubation Success Rate; Propofol Adverse Reaction
Keywords: Cecal intubation; Psychomotor recovery; Procedural sedation; Colonoscopy
MeSH Terms: interventions — Propofol; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol withdrawal arm (Experimental): This group will undergo withholding of the propofol sedation upon intubating the cecum during the colonoscopy.
  Interventions: Drug: propofol (drug)
- Propofol continuation arm (No Intervention): This group will not undergo propofol sedation stoppage upon intubating the cecum during the colonoscopy, and will continue receiving continuous intravenous propofol until the full withdrawal of the colonoscope.

INTERVENTIONS:
Drug: propofol (drug) — Withholding the continuous propofol intravenous drip upon intubating the cecum during the colonoscopy.
  Arms: Propofol withdrawal arm

SUMMARY:
This study investigates whether discontinuing the continuous intravenous infusion of propofol immediately after cecal intubation would reduce the patient's recovery time without compromising their comfort or convenience. It would also reduce procedural costs and the risk of medical hazards due to potentially excessive sedation.

DETAILED DESCRIPTION:
Colonoscopy is usually conducted after inducing depression in the patient's level of consciousness through sedation, ranging from minimal anxiolysis to general anesthesia, to establish relief from potential anxiety, discomfort, and pain during the procedure; in addition to diminishing the patient's memory of the event and minimizing the risk of adverse events related to agitation. It is traditionally done under endoscopist-directed conscious sedation via the administration of a benzodiazepine and a narcotic. However, anesthesia-assisted sedation has significantly risen for the last decade using almost exclusively propofol continuous intravenous drip, with propofol being a non-analgesic sedating agent marked by its rapid distribution and elimination and stronger sedating effect than the standard regimen, leading to faster induction and recovery from sedation and higher physician and patient satisfaction rates. Several anesthesia techniques were also introduced to ease the visceral pain associated with colonoscopy, such as intravenous lidocaine infusion, low-dose intravenous ketamine, and inhalation of an anesthetic mixture of oxygen with nitrous oxide.

Nevertheless, procedural sedation can induce mild cognitive decline after seemingly full recovery. Padmanabhan and colleagues report a significant decrease in visual attention and psychomotor function from baseline after sedation for colonoscopy. It is recommended by the guidelines for conscious sedation and monitoring during gastrointestinal endoscopy (ASGE, 2003) and the Institute Review of Endoscopic Sedation (AGA, 2008) that patients should be accompanied home by a responsible individual after endoscopic sedation, in addition to be instructed to avoid driving, make legally binding decisions, or operate heavy or potentially harmful machinery. The investigators have recently shown that an important proportion of patients experience periods of general anesthesia and/or a deep hypnotic state during endoscopy.

Prolonged systemic anesthesia is noted to increase the risk for serious complications in colonoscopy patients, either hemodynamically or psychomotorly. Additionally, Wernli and colleagues showed that the overall risk of complications after colonoscopy within 30 days increases when individuals receive anesthesia services, namely, the increased risk of perforation, abdominal pain, and stroke. Thus, minimizing the time systemic anesthesia is administered to the patient as possible during the procedure will likely reduce its potential side effects.

The withdrawal time following cecal intubation is quite controversial and operator-dependent. However, it is recommended to be between 6 and 9 minutes. Thus, withholding anesthetic agents during this phase might be beneficial. It would reduce the patient's exposure to anesthesia without causing any significant under-sedation until the near end of the procedure. At the same time, this intervention may accelerate the patient's post-procedure psychomotor recovery by terminating systemic sedation at an earlier checkpoint. Moreover, Adenoma detection rate (ADR), which refers to the rate of detecting colonic adenomas, is typically assessed during the withdrawal of the scope after cecal intubation. It is well known that this rate is influenced by the withdrawal time, meaning the duration the colonoscopist spends withdrawing the scope from the patient. Early discontinuation of anesthesia could limit the time available for the colonoscopist to detect adenomas during withdrawal, making it a significant outcome to evaluate after each colonoscopy.

This study explores whether discontinuing the continuous intravenous infusion of propofol directly following cecal intubation would shorten the patient's recovery time without affecting his comfort or convenience. It would also reduce procedural costs and the risk of medical hazards due to potentially excessive sedation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years.
* Scheduled ambulatory elective screening or surveillance colonoscopy under MAC.

Exclusion Criteria:

* Medical contraindication to anesthesia (i.e., respiratory/cardiac/neurologic compromise, known allergy or adverse reaction to propofol, midazolam, lidocaine, or opiates, …)
* History of ischemic or hemorrhagic cerebrovascular accident.
* Baseline cognitive dysfunction (impaired memory, attention deficit, language disorders, …) - in other words, any dysfunction that prevents the subject from understanding the study protocol and/or completing the requested tests and assessments (e.g., playing the minigames, …)
* Use of more than one psychoactive drug.
* History of partial colectomy.
* Unable to give consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time to psychomotor recovery after the completion of the colonoscopy | From enrollment until 24 hours after finishing the colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- The American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Mokahal A, Daher HB, Yamout R, Hoshaimi N, Ayoub C, Shaib Y, et al. Randomized controlled trial of procedural sequence for same-day bidirectional endoscopy under monitored anesthesia care (RECoVER Trial). iGIE. 2023;2(3):282-91.
- [Background] Bou Daher H, El Mokahal A, Ibrahim MA, Yamout R, Hochaimi N, Ayoub C, et al. General anesthesia and/or deep hypnotic state in propofol-based conscious sedation for endoscopy. iGIE. 2024;3(2):286-92.
- [Background] ASGE Standards of Practice Committee; Early DS, Lightdale JR, Vargo JJ 2nd, Acosta RD, Chandrasekhara V, Chathadi KV, Evans JA, Fisher DA, Fonkalsrud L, Hwang JH, Khashab MA, Muthusamy VR, Pasha SF, Saltzman JR, Shergill AK, Cash BD, DeWitt JM. Guidelines for sedation and anesthesia in GI endoscopy. Gastrointest Endosc. 2018 Feb;87(2):327-337. doi: 10.1016/j.gie.2017.07.018. Epub 2018 Jan 3. No abstract available. PMID 29306520